CLINICAL TRIAL: NCT04166409
Title: A Phase 3 Randomized Non-Inferiority Study of Carboplatin and Vincristine Versus Selumetinib (NSC# 748727) in Newly Diagnosed or Previously Untreated Low-Grade Glioma (LGG) Not Associated With BRAFV600E Mutations or Systemic Neurofibromatosis Type 1 (NF1)
Brief Title: A Study of the Drugs Selumetinib vs. Carboplatin and Vincristine in Patients With Low-Grade Glioma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-07600; NCI-2019-07600 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACNS1833 (Other: Children's Oncology Group); ACNS1833 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2019-11-15; First posted 2019-11-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Low Grade Astrocytoma; Low Grade Glioma; Metastatic Low Grade Astrocytoma; Metastatic Low Grade Glioma; WHO Grade 1 Glioma; WHO Grade 2 Glioma
MeSH Terms: interventions — Specimen Handling; Carboplatin; Magnetic Resonance Spectroscopy; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (vincristine sulfate, carboplatin) (Active Comparator): INDUCTION: Patients receive vincristine sulfate IV on days 1, 8, 15, 22, 29, 36, 43, 50, 57, and 64, and carboplatin IV over 60 minutes on days 1, 8, 15, 22, 43, 50, 57, and 64 in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood and MRI throughout the trial.
  MAINTENANCE: Patients receive vincristine sulfate IV on days 1, 8, and 15, and carboplatin IV over 60 minutes on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 42 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood and MRI throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Drug: Vincristine Sulfate
- Arm II (selumetinib sulfate) (Experimental): Patients receive selumetinib sulfate PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for up to 27 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO at baseline and undergo collection of blood and MRI throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Drug: Selumetinib Sulfate

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm I (vincristine sulfate, carboplatin)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
  Arms: Arm II (selumetinib sulfate)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Questionnaire Administration — Ancillary studies
Drug: Selumetinib Sulfate — Given PO
  Other Names: AZD-6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulphate; Koselugo; Selumetinib Sulphate
  Arms: Arm II (selumetinib sulfate)
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: Arm I (vincristine sulfate, carboplatin)

SUMMARY:
This phase III trial compares the effect of selumetinib versus the standard of care treatment with carboplatin and vincristine (CV) in treating patients with newly diagnosed or previously untreated low-grade glioma (LGG) that does not have a genetic abnormality called BRAFV600E mutation and is not associated with systemic neurofibromatosis type 1. Selumetinib works by blocking some of the enzymes needed for cell growth and may kill tumor cells. Carboplatin is in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of tumor cells. Vincristine is in a class of medications called vinca alkaloids. It works by stopping tumor cells from growing and dividing and may kill them. The overall goal of this study is to see if selumetinib works just as well as the standard treatment of CV for patients with LGG. Another goal of this study is to compare the effects of selumetinib versus CV in subjects with LGG to find out which is better. Additionally, this trial will also examine if treatment with selumetinib improves the quality of life for subjects who take it.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate that the efficacy of treatment with selumetinib as measured by event-free survival (EFS) is non-inferior compared to treatment with carboplatin/vincristine (CV) in previously-untreated low-grade glioma (LGG) not associated with BRAFV600E mutations or systemic neurofibromatosis type 1 (NF1).

SECONDARY OBJECTIVES:

I. To estimate tumor response rates to each regimen of chemotherapy. II. To evaluate visual acuity (VA) outcomes utilizing Teller Acuity Cards (TAC) and HOTV letter acuity testing in previously-untreated optic pathway gliomas (OPGs).

III. To describe the improvement in motor function as measured by the Vineland Scale in children with previously-untreated LGG that have motor deficits at enrollment.

IV. To estimate the difference in EFS and tumor response rate between BRAF rearranged and non-BRAF rearranged patients treated on each chemotherapy regimen.

V. To prospectively evaluate the quality of life of children with LGG not associated with BRAFV600E or systemic NF1 treated with either CV or selumetinib.

VI. To prospectively evaluate the cognitive, social, emotional, and behavioral functioning of children with LGG not associated with BRAFV600E or systemic NF1 treated with either CV or selumetinib.

EXPLORATORY OBJECTIVE:

I. To obtain paired blood and tumor specimens for future biology studies as well as data from Molecular Characterization Initiative (MCI) testing, to correlate genomic drivers to efficacy outcomes.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I:

INDUCTION: Patients receive vincristine sulfate intravenously (IV) on days 1, 8, 15, 22, 29, 36, 43, 50, 57, and 64, and carboplatin IV over 60 minutes on days 1, 8, 15, 22, 43, 50, 57, and 64 in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood and magnetic resonance imaging (MRI) throughout the trial.

MAINTENANCE: Patients receive vincristine sulfate IV on days 1, 8, and 15, and carboplatin IV over 60 minutes on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 42 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood and MRI throughout the trial.

ARM II: Patients receive selumetinib sulfate orally (PO) twice daily (BID) on days 1-28 of each cycle. Cycles repeat every 28 days for up to 27 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo echocardiography (ECHO) at baseline and undergo collection of blood and MRI throughout the trial.

After completion of study treatment, patients are followed up every 3 months for year 1, every 6 months for years 2-3, and then annually for years 4-10.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >= 2 years and =< 21 years at the time of enrollment
* Patients must have a body surface area (BSA) of >= 0.5 m^2 at enrollment
* Patients must have non-neurofibromatosis type 1 (non-NF1) low-grade glioma (LGG) without a BRAFV600E mutation as confirmed by Rapid Central Pathology and Molecular Screening Reviews performed on APEC14B1 (NCT02402244) Childhood Cancer Data Initiative (CCDI)-MCI, or accepted Clinical Laboratory Improvement Act (CLIA)-certified test and that has not been treated with any modality besides surgery. Note: Patients may be newly-diagnosed OR previously diagnosed, and there is no required time frame between biopsy/surgery and treatment initiation.

  * Patients with residual tumor after resection or progressive tumor after initial diagnosis (with or without surgery) who have not received treatment (chemotherapy and/or radiation) are eligible
  * Patients must have two-dimensional measurable tumor >= 1 cm^2 to be eligible
  * Patients with ependymoma are not eligible
* Eligible histologies will include all tumors considered low-grade glioma or low-grade astrocytoma (World Health Organization [WHO] grade I and II) by 5th edition WHO classification of central nervous system (CNS) tumors with the exception of subependymal giant cell astrocytoma
* Patients with metastatic disease or multiple independent primary LGG are eligible
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 OR a serum creatinine based on age/sex as follows (performed within 7 days prior to enrollment):

  * Age: Maximum Serum Creatinine (mg/dL)
  * 2 to < 6 years: 0.8 mg/dL (male); 0.8 mg/dL (female)
  * 6 to < 10 years: 1 mg/dL (male); 1 mg/dL (female)
  * 10 to < 13 years: 1.2 mg/dL (male); 1.2 mg/dL (female)
  * 13 to < 16 years: 1.5 mg/dL (male); 1.4 mg/dL (female)
  * >= 16 years: 1.7 mg/dL (male); 1.4 mg/dL (female)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age (performed within 7 days prior to enrollment) (children with a diagnosis of Gilbert's syndrome will be allowed on study regardless of their total and indirect [unconjugated] bilirubin levels as long as their direct [conjugated] bilirubin is < 3.1 mg/dL)
* Serum glutamic pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L (performed within 7 days prior to enrollment). For the purpose of this study, the ULN for SGPT is 45 U/L
* Albumin >= 2 g/dL (performed within 7 days prior to enrollment)
* Left ventricular ejection fraction (LVEF) >= 53% (or institutional normal; if the LVEF result is given as a range of values, then the upper value of the range will be used) by echocardiogram (performed within 4 weeks prior to enrollment)
* Corrected QT (QTc) interval =< 450 msec by electrocardiography (EKG) (performed within 4 weeks prior to enrollment)
* Absolute neutrophil count >= 1,000/uL (unsupported) (performed within 7 days prior to enrollment)
* Platelets >= 100,000/uL (unsupported) (performed within 7 days prior to enrollment)
* Hemoglobin >= 8 g/dL (may be supported) (performed within 7 days prior to enrollment)
* Patients with a known seizure disorder must be stable and must not have experienced a significant increase in seizure frequency within 2 weeks prior to enrollment
* Patients 2-17 years of age must have a blood pressure that is =< 95th percentile for age, height, and sex at the time of enrollment (with or without the use of anti-hypertensive medications)
* Patients >= 18 years of age must have a blood pressure =< 130/80 mmHg at the time of enrollment (with or without the use of anti-hypertensive medications)
* Note for patients of all ages: Adequate blood pressure can be achieved using medication for the treatment of hypertension
* All patients must have ophthalmology toxicity assessments performed within 8 weeks prior to enrollment
* For all patients, an MRI of the brain (with orbital cuts for optic pathway tumors) and/or spine (depending on the site(s) of primary disease) with and without contrast must be performed within 8 weeks prior to enrollment
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1, or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Patients must have the ability to swallow whole capsules
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met
* All patients have signed an appropriate consent form and Health Insurance Portability and Accountability Act (HIPAA) authorization form (if applicable)
* All patients have been consented and enrolled on APEC14B1 (NCT02402244) Part A for Pre-Enrollment Eligibility Screening for ACNS1833

Exclusion Criteria:

* Patients must not have received any prior tumor-directed therapy including chemotherapy, radiation therapy, immunotherapy, or bone marrow transplant. Prior surgical intervention (with the exclusion of laser interstitial thermal therapy [LITT]) is permitted
* Patients with a concurrent malignancy or history of treatment (other than surgery) for another tumor within the last year are ineligible
* Patients with diffuse intrinsic pontine tumors as seen on MRI (> 2/3 of pons involvement on imaging) are not eligible even if biopsy reveals grade I/II histology
* Patients may not be receiving any other investigational agents
* Patients with any serious medical or psychiatric illness/condition, including substance use disorders or ophthalmological conditions, likely in the judgment of the investigator to interfere or limit compliance with study requirements/treatment
* Patients who, in the opinion of the investigator, are not able to comply with the study procedures are not eligible
* Female patients who are pregnant are not eligible since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential
* Lactating females who plan to breastfeed their infants are not eligible
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation and for 1 week after stopping study therapy are not eligible.

  * Note: Women study participants of child-bearing potential must use acceptable contraception during the study and for 1 week (7 days) after the last dose of selumetinib. Men study participants with sexual partners who are pregnant or who are of child-bearing potential must use acceptable contraception during the study and for 1 week (7 days) after the last dose of study agent. Acceptable contraception includes implants, injectables, or oral contraceptives (all combined with barrier methods), some intrauterine devices (IUDs), vasectomy or abstinence
* Known genetic disorder that increases risk for coronary artery disease. Note: The presence of dyslipidemia in a family with a history of myocardial infarction is not in itself an exclusion unless there is a known genetic disorder documented
* Symptomatic heart failure
* New York Health Association (NYHA) class II-IV prior or current cardiomyopathy
* Severe valvular heart disease
* History of atrial fibrillation
* Current or past history of central serous retinopathy
* Current or past history of retinal vein occlusion or retinal detachment
* Patients with uncontrolled glaucoma

  * If checking pressure is clinically indicated, patients with intraocular pressure (IOP) > 22 mmHg or ULN adjusted by age are not eligible
* Supplementation with vitamin E greater than 100% of the daily recommended dose. Any multivitamin containing vitamin E must be stopped prior to study enrollment even if less than 100% of the daily recommended dosing for vitamin E
* Surgery within 2 weeks prior to enrollment, with the exception of surgical biopsy, placement of a vascular access device or cerebral spinal fluid (CSF) diverting procedure such as endoscopic third ventriculostomy (ETV) and ventriculoperitoneal (VP) shunt.

  * Note: Patients must have healed from any prior surgery
* Patients who have an uncontrolled infection are not eligible

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Up to 10 years from date of randomization
  The Kaplan-Meier method will be used to estimate EFS which is defined as the interval from randomization to first occurrence of clinical or radiographic disease progression, disease recurrence, second malignant neoplasm, or death from any cause, or to the date of last follow-up. Estimates with 95% confidence intervals will be reported by treatment arm. The hazard ratio with a confidence interval will also be reported to compare treatment arms based on a Cox proportional hazards model stratified by BRAF status, tumor location and size of residual tumor. Will also provide outcome estimates and their associated confidence intervals by sex, race and ethnicity, as descriptive summaries of outcome.

SECONDARY OUTCOMES:
Radiographic tumor response rate | Up to 10 years
  Percentages of patients with responses (complete or partial response) will be reported by treatment arm with 95% confidence intervals. The result of an exact binomial test to test for the difference in response rates between treatment arm will also be reported. Will also provide outcome estimates and their associated confidence intervals by sex, race and ethnicity, as descriptive summaries of outcome.
Overall survival (OS) | Up to 10 years from date of randomization
  The Kaplan-Meier method will be used to estimate OS by treatment arm, defined as the interval from randomization to death from any cause, or to the date of last follow-up. Estimates with confidence intervals will be reported by treatment arm. Will also provide outcome estimates and their associated confidence intervals by sex, race and ethnicity, as descriptive summaries of outcome.
Number of patients who experience an improvement in visual acuity (VA) | After the first 12 months of treatment
  Numbers of patients that show improvement in VA after 12 months of treatment will be reported by treatment arm. Patients with at least 1 impaired eye are evaluable. In a patient with a unilateral optic nerve glioma, only the affected eye is considered. In patients with bilateral visual impairment, if VA improves in 1 eye but worsens in the other, the patient will be coded as a treatment failure, whereas if 1 eye improves and the other is at least stable, the patient will be coded as a success.
Change in motor function | After 48 weeks of therapy
  Motor function is measured using the Vineland-3 Motor Scale. Only patients with motor function deficits at baseline are included. Magnitudes of change from baseline between the 2 treatment arms and provide a 90% 2-sided confidence interval for this difference.
Change in quality of life (QOL) | Baseline and 9 months after treatment initiation
  QOL will be measured using the PedsQL Total Scale Score as measured from the validated PedsQL Generic Module (for children 2-21 years old). Mean differences in the total scale score between 9 months and baseline will be reported by treatment arm. The results of 2-sample t-test comparing differences in the QOL scores between the 2 arms will also be reported. If change scores do not follow normal distributions, non-parametric alternatives may be employed for analysis.
Processing speed function | Up to 9 months post-treatment initiation
  Measured by Wechsler Processing Speed Index (standard score). Scores at 9 months will be summarized by treatment arm and reported as means (with standard deviations) or medians (with ranges) depending on the data distribution.
Change in executive function | Baseline and 9-months
  Executive function will be measured by the Behavior Rating Inventory of Executive Function, Second Edition BRIEF Cognitive Regulation Index (CRI). Summary statistics for the differences in scores from baseline to 9 months will be reported by treatment arm.

OTHER OUTCOMES:
Change in QOL scores over time | At baseline, 9 months, 30 months, and 60 months after treatment initiation
  QOL scores for each domain of the PedsQL Generic module will be summarized by timepoint (4 timepoints) and treatment arm. Mean QOL scores will be reported with standard deviations. If scores do not follow normal distributions, medians and ranges will be reported instead.
Change in neurocognitive functioning scores over time | At baseline, 9 months, 30 months, and 60 months after treatment initiation
  Neurocognitive functioning scores for each index/scale of the Behavior Rating Inventory of Executive Function, Second Edition/Preschool Version/Adult will be summarized by timepoint (4 timepoints) and treatment arm. Mean scores will be reported with standard deviations. If scores do not follow normal distributions, medians and ranges will be reported instead.
EFS by sex | Up to 10 years from date of randomization
  Estimates of treatment effect and the corresponding 95% confidence intervals will be provided by sex.
EFS by race | Up to 10 years from date of randomization
  Estimates of treatment effect and the corresponding 95% confidence intervals will be provided by race.
EFS by ethnicity | Up to 10 years from date of randomization
  Estimates of treatment effect and the corresponding 95% confidence intervals will be provided by ethnicity.
OS by sex | Up to 10 years from date of randomization
  Estimates of treatment effect and the corresponding 95% confidence intervals will be provided by sex.
OS by race | Up to 10 years from date of randomization
  Estimates of treatment effect and the corresponding 95% confidence intervals will be provided by race.
OS by ethnicity | Up to 10 years from date of randomization
  Estimates of treatment effect and the corresponding 95% confidence intervals will be provided by ethnicity.
Neurocognitive outcomes by sex | Up to 10 years from date of randomization
  Estimates of treatment effect and the corresponding 95% confidence intervals will be provided by sex.
Neurocognitive outcomes by race | Up to 10 years from date of randomization
  Estimates of treatment effect and the corresponding 95% confidence intervals will be provided by race.
Neurocognitive outcomes by ethnicity | Up to 10 years from date of randomization
  Estimates of treatment effect and the corresponding 95% confidence intervals will be provided by ethnicity.
QOL by sex | Up to 10 years from date of randomization
  Estimates of treatment effect and the corresponding 95% confidence intervals will be provided by sex.
QOL by race | Up to 10 years from date of randomization
  Estimates of treatment effect and the corresponding 95% confidence intervals will be provided by race.
QOL by ethnicity | Up to 10 years from date of randomization
  Estimates of treatment effect and the corresponding 95% confidence intervals will be provided by ethnicity.

CONTACTS AND LOCATIONS:
Overall Officials: Peter M de Blank, Principal Investigator — Children's Oncology Group
Locations (132):
- United States (124):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (7):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- HIMA San Pablo Oncologic Hospital, Caguas, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Bergqvist C, Wolkenstein P. MEK inhibitors in RASopathies. Curr Opin Oncol. 2021 Mar 1;33(2):110-119. doi: 10.1097/CCO.0000000000000711. PMID 33395032
- [Derived] Arnold A, Rodriguez F, Eberhart CG, Raabe EH. Response to letter to the editor: "All models are wrong; some models are useful". Neuro Oncol. 2020 Sep 29;22(9):1406-1407. doi: 10.1093/neuonc/noaa137. No abstract available. PMID 32597469